CLINICAL TRIAL: NCT07316309
Title: A Prospective Study of [18F]AlF-NOTA-QHY-04 PET/CT for Predicting Outcome in Patients With Limited-Stage Small Cell Lung Cancer Treated With Concurrent Chemoradiotherapy
Brief Title: CXCR4 PET/CT for Predicting Outcome in Limited-Stage Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jie Liu, Principal Investigator, Shandong Cancer Hospital and Institute
Other Study IDs: QHY04-LS-SCLC-01
Record Dates: First submitted 2025-12-18; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Limited-Stage Small Cell Lung Cancer Cohort: Patients with histologically confirmed limited-stage small cell lung cancer who were enrolled prospectively and received standard-of-care treatment according to institutional protocols.

SUMMARY:
This prospective observational study aims to evaluate the clinical value of CXCR4-targeted PET/CT imaging in patients with limited-stage small cell lung cancer (LS-SCLC).

Patients diagnosed with LS-SCLC at Shandong Cancer Hospital and Institute underwent [18F]AlF-NOTA-QHY-04 PET/CT imaging before receiving standard concurrent chemoradiotherapy. Imaging findings were analyzed and correlated with clinical outcomes, including progression-free survival, to explore the potential role of CXCR4 PET/CT as a prognostic imaging biomarker.

The results of this study may help improve risk stratification and outcome prediction in patients with limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
This was a single-center, prospective observational study conducted at Shandong Cancer Hospital and Institute to investigate the prognostic value of CXCR4-targeted PET/CT imaging in patients with limited-stage small cell lung cancer (LS-SCLC).

Eligible patients with histologically confirmed LS-SCLC underwent [18F]AlF-NOTA-QHY-04 PET/CT imaging prior to standard concurrent chemoradiotherapy. PET/CT parameters reflecting CXCR4 expression were measured and analyzed.

Patients were subsequently followed up according to routine clinical practice. Clinical outcomes, including progression-free survival and overall survival, were recorded during follow-up. The association between baseline CXCR4 PET/CT imaging findings and clinical outcomes was evaluated to explore the potential role of CXCR4-targeted PET/CT as a prognostic imaging biomarker in LS-SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed limited-stage small cell lung cancer (T1-4N0-3M0) according to the AJCC TNM 8th edition.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Presence of measurable disease according to RECIST version 1.1.
* Newly diagnosed patients who had not received any prior anticancer treatment.
* Underwent baseline [18F]AlF-NOTA-QHY-04 PET/CT imaging prior to treatment.

Exclusion Criteria:

* Presence of autoimmune diseases or active comorbid infections.
* Pregnancy or breastfeeding.
* Unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with newly diagnosed, histopathologically confirmed limited-stage small cell lung cancer who underwent baseline [18F]AlF-NOTA-QHY-04 PET/CT imaging prior to concurrent chemoradiotherapy at Shandong Cancer Hospital and Institute.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Progression Status at 6 Months After Completion of Concurrent Chemoradiotherapy (CCRT) | 6 months after completion of concurrent chemoradiotherapy (CCRT)
  Progression status assessed at 6 months after completion of concurrent chemoradiotherapy (CCRT) using imaging evaluation according to RECIST version 1.1. Participants were classified as having progression (Progressors) or no progression (Non-progressors).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From date of enrollment until the date of first documented progression (per RECIST version 1.1) or date of death from any cause, whichever came first, assessed up to 36 months
  Progression-free survival, defined as the time from study enrollment to disease progression (per RECIST version 1.1) or death from any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Liu, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.